CLINICAL TRIAL: NCT01579149
Title: A Phase 1, Randomized, Single-center, Single-dose, Double-blind, Placebo-controlled Pharmacokinetic, Safety, and Pharmacodynamic Study of Subcutaneous Injection of 160 μg/kg, 240 μg/kg, and 400 μg/kg Plerixafor in Healthy Adult Volunteers of Japanese Descent
Brief Title: A Phase I Dose Escalation Study of Plerixafor in Healthy Subjects of Japanese Descent
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOZ24211
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — plerixafor

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- plerixafor (Experimental): Single subcutaneous (SC) dose of plerixafor (160 μg/kg, 240 μg/kg, or 400 μg/kg)
  Interventions: Drug: plerixafor
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: plerixafor — Single subcutaneous (SC) dose of plerixafor (160 μg/kg, 240 μg/kg, or 400 μg/kg),
  Arms: plerixafor
Drug: Placebo — Single subcutaneous (SC) dose of placebo
  Arms: Placebo

SUMMARY:
The primary objective is to assess the pharmacokinetics of 3 dose levels of plerixafor injection (160 μg/kg, 240 μg/kg, and 400 μg/kg) in healthy adult subjects of Japanese descent. Three cohorts of subjects will be enrolled. Approximately 8 subjects will be enrolled in each cohort, 6 subjects who will receive a single subcutaneous (SC) dose of plerixafor (160 μg/kg, 240 μg/kg, or 400 μg/kg), and 2 subjects who will receive a single SC dose of placebo. The lowest dose-level cohort (plerixafor 160 μg/kg) will be fully enrolled first, followed by the next highest dose-level cohort (plerixafor 240 μg/kg), and finally the highest dose-level cohort (plerixafor 400 μg/kg), provided safety criteria for dose escalation are met.

DETAILED DESCRIPTION:
Screening will occur within 28 days prior to dosing. Dosing will occur on Day 1 of each cohort. Subjects will remain at the study center from Day -1 until discharge approximately 24 hours after dosing (Day 2) for pharmacokinetic, safety, and pharmacodynamic assessments; however, all subjects who receive any investigational product, including any subjects who prematurely withdraw from the study, will remain at the study center for a minimum of 4 hours after dosing. A 15-day follow-up visit will be conducted 15 to 20 days postdose. The study will be considered completed for a subject at the time he/she completes the 15-day follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects of Japanese descent, i.e., the subject was born in Japan and has lived outside of Japan for <10 years, and the subject's biological parents and grandparents are fully Japanese and were born in Japan.
* Subjects with body weight <95.0 kg if male, <85.0 kg if female, and <175% of ideal body weight (IDW)
* The subject has estimated creatinine clearance 50 mL/min or higher as determined by the Cockcroft-Gault formula.
* The subject's serum creatinine, alkaline phosphatase, hepatic enzymes (aspartate aminotransferase [AST], alanine aminotransferase [ALT]), and total bilirubin (unless the subject has documented Gilbert syndrome) should not exceed the upper laboratory normal limit. Other biochemistry, hematology, and urinalysis laboratory parameters must not exceed National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 1.
* The subject is negative for HIV, active hepatitis B, and active hepatitis C.
* The subject refrained from consuming alcohol for 48 hours prior to Day 1 and agrees to refrain from alcohol consumption through discharge from the center and 24 hours prior to the follow-up visit (Day 15 [+5 days]).
* Female subjects of child-bearing potential and male subjects with partners of child-bearing potential agree to use an effective means of birth control while on study therapy and for a minimum of 1 month following final study visit. Effective birth control includes: (a) birth control pills, depot progesterone, or an intrauterine device plus one barrier method; or (b) 2 barrier methods. Effective barrier methods are male and female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). For subjects using a hormonal contraceptive method, information about any interaction of plerixafor with hormonal contraceptives is not known.
* The subject has given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

* History of clinically significant cardiac disorders, pulmonary disorders, malignancy, or other major medical issues that, in the view of the Investigator, renders the subject at high risk from treatment complications.
* Known allergy or sensitivity to plerixafor.
* Blood donation within 30 days prior to Day 1.
* Active infection, including unexplained fever (temperature >38.1ºC) or antibiotic and/or antiviral therapy within 7 days prior to Day 1.
* Abnormal electrocardiogram (ECG) with clinically significant conduction (heart block; or QTc >430 ms [males] or QTc >450 ms [females]) or rhythm disturbance (ventricular arrhythmias) within 1 year prior to Day 1 that, in the opinion of the Investigator, warrants exclusion of the subject from the study.
* History or known current alcohol, narcotic, or illicit drug abuse within the past 5 years.
* If female, pregnant (defined as positive serum β-HCG test) or lactating.
* Any medication, including over-the-counter medications and/or alternative medication (eg, dietary, herbal, botanical, or homeopathic supplements), within 7 days prior to Day 1, with the exception of hormonal birth control.
* Blood transfusion in the 30 days prior to Day 1.
* The subject does not tolerate venipuncture.
* In the opinion of the Investigator, subject is unable to adhere to the requirements of the study.
* The subject previously received investigational therapy within 4 weeks of Day 1 or within 6 weeks of Day 1 in the case of a long-acting agent (half-life >14 days) such as an antibody, is currently enrolled in another investigational protocol, or plans to receive any other investigational product at any time during the course of this study up to the time of the final follow-up visit.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics as measured by maximum observed concentration (Cmax) | Pre-dose to 24 hours post-dose
Pharmacokinetics as measured by time to maximum concentration (Tmax) | Pre-dose to 24 hours post-dose
• Pharmacokinetics as measured by area under the concentration-time curve (AUC) from Time 0 to 24 hours post-dose | Pre-dose to 24 hours post-dose
Pharmacokinetics as measured by terminal half-life (t1/2) | Pre-dose to 24 hours post-dose
Pharmacokinetics as measured by apparent volume of distribution (Vz/F) | Pre-dose to 24 hours post-dose
Pharmacokinetics as measured by apparent total systemic clearance (CL/F) | Pre-dose to 24 hours post-dose

SECONDARY OUTCOMES:
Safety as measured by incidence of treatment-emergent adverse events (AEs) and serious adverse events (SAEs) | From the administration of study drug and up to 15 day follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Honolulu, Hawaii, United States